CLINICAL TRIAL: NCT01459159
Title: Phase 2b Study of Oral Ezatiostat Hydrochloride (Telintra®) in Patients With Low to Intermediate-1 Risk, Non-Deletion 5q Myelodysplastic Syndrome
Brief Title: Study of (Telintra®) in Non-Del(5q) Myelodysplastic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study TLK199.2108 was terminated for business reasons.
Sponsor: Telik (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLK199.2108
Record Dates: First submitted 2011-10-11; First posted 2011-10-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: Hematology; MDS; Myelodysplastic Syndrome; Low risk MDS; Int-1 risk MDS; Transfusion dependence; Telintra; ezatiostat; ezatiostat hydrochloride; TLK199; Glutathione; Glutathione analog; Glutathione Transferase; Glutathione Transferase P1-1 inhibitor; GST P1-1 inhibitor; Apoptosis; Differentiation; Enzyme inhibitor; non-del (5q); non-deletion 5q
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — gamma-Glu-S-BzCys-PhGly diethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ezatiostat hydrochloride (Telintra®) — Three weeks of treatment with ezatiostat at 2000 mg per day in divided doses followed by a one week rest period in four-week treatment cycles.
  Other Names: Telintra; Telintra Tablets; Oral Telintra; ezatiostat; ezatiostat hydrochloride; oral ezatiostat

SUMMARY:
This is a multicenter, single arm open label Phase 2b Study of oral ezatiostat (Telintra®) in Patients who are RBC tranfusion dependent, Low to INT-1 IPSS risk, non-del (5q) Myelodysplastic Syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria:

* Primary or de Novo MDS
* Low to Intermediate-1 IPSS risk of MDS
* ECOG performance score of 0 or 1
* Documentation of significant anemia with or without additional cytopenia
* Adequate kidney and liver function
* Patients must have discontinued hematopoietic growth factors at least 3 weeks prior to study entry

Exclusion Criteria:

* Deletion of the 5q chromosome [del(5q) MDS]
* Prior allogenic bone marrow transplant for MDS
* Known sensitivity to ezatiostat (injection or oral tablets)
* Prior treatment with hypomethylating agent (HMA) (e.g., azacitadine, decitabine)
* History of MDS IPSS risk score of greater than 1.0
* Pregnant or lactating women
* Any severe concurrent disease, infection or comorbidity that, in the judgement of the investigator, would make the patient inappropriate for study entry
* Oral steroids greater than 10 mg per day. Exceptions: those prescribed for other conditions (such as new adrenal failure, asthma, arthritis) or brief sterioid use (such as tapered dosing for an acute non-MDS condition)
* History of hepatitis B or C, or HIV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Hematologic Improvement-Erythroid (HI-E) rate | At 8 weeks of treatment
  Hematologic Improvement response will be assessed per the IWG MDS response criteria (2006)
Hematologic Improvement-Erythroid (HI-E) rate | At 16 weeks of treatment
  Hematologic Improvement response will be assessed per the IWG MDS response criteria (2006)
Hematologic Improvement-Erythroid (HI-E) rate | At 24 weeks of treatment
  Hematologic Improvement response will be assessed per the IWG MDS response criteria (2006)
Hematologic Improvement-Erythroid (HI-E) rate | At 32 weeks of treatment
  Hematologic Improvement response will be assessed per the IWG MDS response criteria (2006)

SECONDARY OUTCOMES:
RBC Transfusion independence (TI) rate | At 4, 8, 12, 16, 20, 24, 28 & 32 weeks of treatment
Hematologic Improvement-Neutrophil (HI-N) rate | At 8, 16, 24, & 32 weeks of treatment
  Hematologic Improvement response will be assessed per the IWG MDS response criteria (2006)
Hematologic Improvement-Platelet (HI-P) rate | At 8, 16, 24, & 32 weeks of treatment
  Hematologic Improvement response will be assessed per the IWG MDS response criteria (2006)
Unilineage, bilineage, trilineage, and overall HI response rate | 2 years
Cytogenetic response rate | 16 weeks, 48 weeks and at the time of first HI response
Duration of response | 2 years
Safety of ezatiostat in this MDS population | At 4, 8, 12, 16, 20, 24, 28 & 32 weeks of treatment
  Recording and grading of AEs using NCI-CTCAE v4.03
Evaluation of the relationship between HI-E response, gene expression profiling and response-related variables | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gail L Brown, MD, Study Director — Telik
Locations (7):
- United States (7):
  - Bay Area Cancer Research Group, Concord, California
  - University of Colorado, Aurora, Colorado
  - SIU School of Medicine, Simmons Cancer Institute, Springfield, Illinois
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Columbia University, New York, New York
  - The West Clinic, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee